CLINICAL TRIAL: NCT00731133
Title: Open-Label Pilot Study of Disulfiram for Methamphetamine Dependence
Brief Title: Open-Label Disulfiram for Methamphetamine Dependence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5-P50-DA018197-105242; 5P50DA018197 (NIH); DPMCDA
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-01

CONDITIONS: Methamphetamine Dependence
Keywords: disulfiram; methamphetamine dependence; open label
MeSH Terms: interventions — Disulfiram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Disulfiram (Other): Disulfiram at 250 mg daily
  Interventions: Drug: Disulfiram

INTERVENTIONS:
Drug: Disulfiram — 250 mg/day
  Other Names: Antabuse

SUMMARY:
This 8 week, open-label pilot clinical trial will examine the safety and tolerability of disulfiram at 250 mg/day in up to fifteen methamphetamine dependent individuals. After undergoing screening procedures (approximately one week), eligible subjects will enter the study proper attend clinic every weekday during week 1 of the trial in order to receive the disulfiram under observation and complete assessments. Then subjects will receive weekly blister packs of medication and attend clinic thrice weekly during weeks 2-6. During weeks 7-8, subjects no longer take disulfiram, are followed for two weeks, then referred to treatment elsewhere, if desired. Urine samples will be obtained and a disulfiram side-effects checklist will be completed thrice-weekly. Self-reported drug use, craving and mood ratings will be completed weekly. All subjects undergo cognitive behavioral therapy. Adjunctive contingency management procedures will be utilized to enhance retention. The primary outcomes of interest include retention, side-effects, and drug use. Our hypothesis is that disulfiram will be well tolerated in this population.

DETAILED DESCRIPTION:
This 8 week, open-label pilot clinical trial will examine the safety and tolerability of disulfiram at 250 mg/day in up to fifteen methamphetamine dependent individuals. After undergoing screening procedures (approximately one week), eligible subjects will enter the study proper attend clinic every weekday during week 1 of the trial in order to receive the disulfiram under observation and complete assessments. Then subjects will receive weekly blister packs of medication and attend clinic thrice weekly during weeks 2-6. During weeks 7-8, subjects no longer take disulfiram, are followed for two weeks, then referred to treatment elsewhere, if desired. Urine samples will be obtained and a disulfiram side-effects checklist will be completed thrice-weekly. Self-reported drug use, craving and mood ratings will be completed weekly. All subjects undergo cognitive behavioral therapy. Adjunctive contingency management procedures will be utilized to enhance retention. The primary outcomes of interest include retention, side-effects, and drug use. Results of this study will provide initial safety and drug use data for grant applications proposing to examine the clinical efficacy of disulfiram or similar agents to for treating methamphetamine dependence under placebo-controlled, double-blind conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* not currently enrolled in a treatment program
* subjects must have a history of methamphetamine use with recent use confirmed by a positive urine toxicology screen for amphetamines during the month prior to study entry
* subjects must meet DSM-IV criteria for amphetamine dependence as assessed by the substance abuse section of the Structured Clinical Interview for DSM-IV (SCID)
* women of childbearing age must have a negative pregnancy test to enroll in this study, agree to monthly pregnancy testing, and agree to use appropriate forms of birth control for the duration of the study.

Exclusion Criteria:

* current diagnosis of alcohol physical dependence
* significant medical conditions such as abnormal liver function (e.g., laboratory findings on ALT or AST greater than three times normal), active hepatitis, uncontrolled hypertension, a current cardiac condition or high risk of cardiovascular disease (see section c.1), seizure disorders, or another significant underlying medical condition which would contraindicate disulfiram treatment
* meeting DSM-IV psychiatric classifications for schizophrenia, bipolar disorder, or other psychotic disorders
* exhibiting current suicidality or homicidality
* pregnancy or breastfeeding
* current use of a prescribed psychotropic medication (e.g., antidepressants, anxiolytics, antipsychotics, anticonvulsants, etc.) which cannot be discontinued
* current use of medications such as anticoagulants, isoniazid, metronidazole, clotrimazole, and paraldehyde

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Disulfiram
Started | 15
Completed | 5
Not Completed | 10
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Arm/Group | Disulfiram
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.93 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Side Effects Checklist
Description: It consists of 25 items describing side effects specific to disulfiram alone or combined with alcohol or cocaine that are rated on a scale from 0 (not at all) to 4 (very much). Total scores range from 0 (minimum) to 100 (maximum). Data were entered into a mixed model ANOVA in order to determine whether scores significantly changed over time. A slope and standard deviation describing this change over time were generated and used as our outcome measures.
Time Frame: Weekly for six weeks
Population: Those who received more than one dose of disulfiram and/or completed more than one set of assessments during the protocol. Of the 15 participants who entered the study, one participant only attended clinic one day and so data were analyzed for 14 participants.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Disulfiram 250 mg
Number analyzed (Participants) | 14
units on a scale | 9.6515 (2.4750)
Statistical Analysis 1: Comparison: Disulfiram 250 mg; Open-label study testing for change in side-effects ratings over time (i.e., slope); Test type: Superiority or Other; p = 0.05, Mixed Models Analysis; 7,24; Slope = 2.6466, 95% CI 2-sided [.7858 to 4.5073], Standard Error of Mean 0.9016

2. Secondary Outcome: Proportion of Amphetamine-positive Urine Samples
Description: the proportion of urine samples positive for amphetamine. Data were entered into a mixed model ANOVA in order to determine whether scores significantly changed over time. A slope and standard deviation describing this change over time were generated and used as our outcome measures.
Time Frame: thrice weekly for 6 weeks
Population: Only data from participants who received more than one dose of disulfiram were analyzed. Of the 15 participants who entered the study, one participant received only one dose so data from 14 participants were analyzed.
Measure: Least Squares Mean (Standard Deviation); unit: proportion of urines positive for amphet
Arm/Group | Disulfiram 250 mg
Number analyzed (Participants) | 14
proportion of urines positive for amphet | 0.3639 (0.1113)
Statistical Analysis 1: Comparison: Disulfiram 250 mg; Open label study testing changes in amphetamine use over time (i.e., slope); Test type: Superiority or Other; p = 0.05, Mixed Models Analysis; 7,24; Slope = -0.3730, 95% CI 2-sided [-0.8075 to 0.06150], Standard Error of Mean 0.2196

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Disulfiram
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 7/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Disulfiram (N=15)
Nausea/Vomitting (Gastrointestinal disorders) | 4/14 (5)
Headache (Nervous system disorders) | 2/14 (2)
Increased blood pressure (Cardiac disorders) | 1/14 (1)
Confusion (Psychiatric disorders) | 1/14 (1)
Sleepiness (General disorders) | 1/14 (1)
Stomach Bloating (Gastrointestinal disorders) | 1/14 (1)
Blurry vision (Nervous system disorders) | 1/14 (1)
Dizziness (General disorders) | 1/14 (1)
Anxiety/Racing Heart (Psychiatric disorders) | 1/14 (1)
Metallic Taste (Gastrointestinal disorders) | 1/14 (1)

LIMITATIONS AND CAVEATS:
Large dropout so few participants had data throughout the trial. No control group so cannot determine whether side effects were related to disulfiram or an artifact of participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes